CLINICAL TRIAL: NCT05120635
Title: Intracranial Neurophysiological Signatures of Fear and Anxiety in Humans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); VA Greater Los Angeles Healthcare System (U.S. Federal Agency); NeuroPace (Industry); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: PRO00118015; R01MH124761 (NIH); Pro00117931 (Other: Duke University)
Record Dates: First submitted 2021-10-04; First posted 2021-11-15 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-09

CONDITIONS: Fear; GAD; Emotional Memory; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EMU Participants (Other): Subjects participating in the study at the Epilepsy Monitoring Unity (EMU).
  Interventions: Device: Deep Brain Stimulation; Behavioral: Virtual and augmented reality tasks
- RNS Participants (Other): Subjects with RNS implants.
  Interventions: Device: Deep Brain Stimulation; Behavioral: Virtual and augmented reality tasks

INTERVENTIONS:
Device: Deep Brain Stimulation — Deep brain stimulation will be used
Behavioral: Virtual and augmented reality tasks — Virtual and augmented reality tasks will be used.

SUMMARY:
Anxiety disorders such as post-traumatic stress disorder (PTSD) and generalized anxiety disorder (GAD) affect a large number of individuals with a significant portion of patients failing to improve with current treatments.

The purpose of this study is to understand the brain mechanisms that produce fear and anxiety in humans. To accomplish this goal, we will measure the brain activity along with the heart rate and skin perspiration of patients while they are completing tasks on a computer. Some of the tasks will also use a virtual reality headset and transport the patient in a video game-like environment. These tasks will expose the participants to various levels of fear-provoking images. Participants with responsive neurostimulation (RNS) implants will be enrolled under Pro00117931 at Duke, but their results for fear and anxiety tasks will be reported under NCT05120635.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Has undergone acute depth or chronic responsive neurostimulation (RNS) electrode placement
* Willing to provide informed consent and participate in the study
* Ability to read and write English fluently

Exclusion Criteria:

* Unwilling to provide informed consent
* Has not undergone acute depth or chronic responsive neurostimulation (RNS) electrode placement
* Pregnant women
* Participants with active psychosis
* Participants with suicidal ideation
* Participants with substance abuse issues

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Physiological change - eye-blinks | during the intervention/behavioral tasks with and without stimulation
  Eye blinks will be measured using an eye tracking device and will be measure in blinks per second.
Physiological change - heart rate variability | during the intervention/behavioral tasks with and without stimulation
  heart rate variability will be measured in milliseconds.
Physiological change - skin conductance | during the intervention/behavioral tasks with and without stimulation
  Skin conductance will be measured in microSiemens.
Neurophysiological activity | during the intervention/behavioral tasks with and without stimulation
  Neurophysiological activity will be measured in Hz

CONTACTS AND LOCATIONS:
Overall Officials: Nanthia Suthana, PhD, Principal Investigator — Duke Health
Locations (2):
- United States (2):
  - University of California Los Angeles, Los Angeles, California
  - Duke University Health System, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No